CLINICAL TRIAL: NCT00380562
Title: Experience Corps Trial: Improving Health of Older Populations Through Generativity
Brief Title: The Baltimore Experience Corps Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Retirement Research Foundation (Other); Abell Foundation (Other); National Institute on Aging (NIA) (NIH); Goldseker Foundation (Unknown); The Harry & Jeanette Weinberg Foundation, Inc. (Other)
Responsible Party: Principal Investigator, George W. Rebok, PhD, Professor, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AG0069; P01AG027735 (NIH)
Record Dates: First submitted 2006-09-25; First posted 2006-09-26 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-09

CONDITIONS: Aging; Generativity
Keywords: Quality of life; Cognitive Functioning; Activities of Daily Living; Disability prevention

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Volunteer (Experimental): High intensity volunteering (15 hours a week or greater) in Baltimore City Schools with children in grades K-3
  Interventions: Behavioral: Experience Corps
- Control (No Intervention): Usual activities

INTERVENTIONS:
Behavioral: Experience Corps — High intensity volunteering (15 hours a week or more) over a two year time period working with children in grades K-3 in Baltimore City Schools. Controls are assigned to usual activities for two years and then offered opportunity to volunteer with children at the end of two year.
  Arms: Volunteer

SUMMARY:
The purpose of this study is to examine the effectiveness of the Experience Corps program in preventing or delaying physical disability in older adults, by studying the effects of volunteerism on physical, social and cognitive well-being.

DETAILED DESCRIPTION:
The Baltimore Experience Corps Study is a randomized, controlled, community-based trial of the effectiveness of Experience Corps (EC) to determine if participation for adults 60 years and older, over two years of follow-up, results in better outcomes in the EC versus control arm in terms of mobility, strength, balance, and cognitive functioning.

The Experience Corps is a community-based model for health promotion for older adults embedded within a social engagement program. The program places older adult volunteers in meaningful roles in public elementary schools, bringing the time, experience, and wisdom of older adults to bear in improving academic and behavioral outcomes of children. The Experience Corps incorporates health promotion preventing disability and dependency associated with aging, into new, generative roles for older adults.

This program was initially designed by Dr. Linda Fried of this application, along with Marc Freedman of Civic Ventures, Inc. It has gone through two national demonstrations, neither of which evaluated the impact on older adults.

ELIGIBILITY:
Inclusion Criteria:

* 60 years or older
* Agree to commit to at least 1 year of participation in the EC and to participate at least 15 hours per week for the full school year, if randomized to the intervention group
* Meet minimum criteria for cognitive functioning necessary to function successfully in a school setting
* Functionally literate, using a nationally recognized and standardized evaluation which provides grade level equivalency in reading and spelling
* Ability to travel to the schools, if randomized to the intervention group
* Agree to accept randomization and to participate in evaluations
* Clearance on the Baltimore city public school's criminal background check, if randomized to intervention group
* Complete training, if randomized to intervention group

Exclusion Criteria:

* Under 60 years of age

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 702 (Actual)
Dates: Start 2006-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Decreased disability in mobility and Instrumental Activities of Daily Living (IADL) | Measured in 4 month intevals from baseline to 24 month
  Walking speed, chair stands, questionnaires related to mobility and activities

SECONDARY OUTCOMES:
Decreased falls | Measured in 4 month intervals from baseline to 24 month
decreased rate of decline in memory | Measured in 4 month intervals from baseline to 24 month
increased, preserved or slowed decline in strength, balance, walking speed, frailty, timed "get up and go", cortical plasticity and executive function and speed and accuracy in objective IADL task performance | Measured in 4 month intervals from baseline to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: George Rebok, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Center on Aging and Health, Baltimore, Maryland, United States

REFERENCES:
- [Background] Fried LP, Carlson MC, Freedman M, Frick KD, Glass TA, Hill J, McGill S, Rebok GW, Seeman T, Tielsch J, Wasik BA, Zeger S. A social model for health promotion for an aging population: initial evidence on the Experience Corps model. J Urban Health. 2004 Mar;81(1):64-78. doi: 10.1093/jurban/jth094. PMID 15047786
- [Background] Frick KD, Carlson MC, Glass TA, McGill S, Rebok GW, Simpson C, Fried LP. Modeled cost-effectiveness of the Experience Corps Baltimore based on a pilot randomized trial. J Urban Health. 2004 Mar;81(1):106-17. doi: 10.1093/jurban/jth097. PMID 15047789
- [Background] Fried LP, Carlson MC, McGill S, Seeman T, Xue QL, Frick K, Tan E, Tanner EK, Barron J, Frangakis C, Piferi R, Martinez I, Gruenewald T, Martin BK, Berry-Vaughn L, Stewart J, Dickersin K, Willging PR, Rebok GW. Experience Corps: a dual trial to promote the health of older adults and children's academic success. Contemp Clin Trials. 2013 Sep;36(1):1-13. doi: 10.1016/j.cct.2013.05.003. Epub 2013 May 13. PMID 23680986
- [Background] Tan EJ, McGill S, Tanner EK, Carlson MC, Rebok GW, Seeman TE, Fried LP. The evolution of an academic-community partnership in the design, implementation, and evaluation of experience corps(R) Baltimore city: a courtship model. Gerontologist. 2014 Apr;54(2):314-21. doi: 10.1093/geront/gnt072. Epub 2013 Jul 25. PMID 23887931
- [Background] Parisi JM, Rebok GW, Seeman TE, Tanner EK, Tan EJ, Fried LP, Xue QL, Frick KD, Carlson MC. Lifestyle Activities in Sociodemographically at-risk Urban, Older Adults Prior to Participation in the Baltimore Experience Corps((R)) Trial. Act Adapt Aging. 2012 Jan 1;36(3):242-260. doi: 10.1080/01924788.2012.702306. Epub 2012 Sep 18. PMID 23144524
- [Background] Parisi JM, Rebok GW, Xue QL, Fried LP, Seeman TE, Tanner EK, Gruenewald TL, Frick KD, Carlson MC. The role of education and intellectual activity on cognition. J Aging Res. 2012;2012:416132. doi: 10.1155/2012/416132. Epub 2012 Aug 9. PMID 22928110
- [Background] Agbedia OO, Varma VR, Seplaki CL, Seeman TE, Fried LP, Li L, Harris GC, Rebok GW, Xue QL, Tan EJ, Tanner E, Parisi JM, McGill S, Carlson MC. Blunted diurnal decline of cortisol among older adults with low socioeconomic status. Ann N Y Acad Sci. 2011 Aug;1231:56-64. doi: 10.1111/j.1749-6632.2011.06151.x. PMID 21884161
- [Background] Tan EJ, Tanner EK, Seeman TE, Xue QL, Rebok GW, Frick KD, Carlson MC, Wang T, Piferi RL, McGill S, Whitfield KE, Fried LP. Marketing public health through older adult volunteering: Experience Corps as a social marketing intervention. Am J Public Health. 2010 Apr;100(4):727-34. doi: 10.2105/AJPH.2009.169151. Epub 2010 Feb 18. PMID 20167888
- [Background] Carlson MC, Erickson KI, Kramer AF, Voss MW, Bolea N, Mielke M, McGill S, Rebok GW, Seeman T, Fried LP. Evidence for neurocognitive plasticity in at-risk older adults: the experience corps program. J Gerontol A Biol Sci Med Sci. 2009 Dec;64(12):1275-82. doi: 10.1093/gerona/glp117. Epub 2009 Aug 19. PMID 19692672
- [Background] Tan EJ, Rebok GW, Yu Q, Frangakis CE, Carlson MC, Wang T, Ricks M, Tanner EK, McGill S, Fried LP. The long-term relationship between high-intensity volunteering and physical activity in older African American women. J Gerontol B Psychol Sci Soc Sci. 2009 Mar;64(2):304-11. doi: 10.1093/geronb/gbn023. Epub 2009 Jan 29. PMID 19181687
- [Background] Carlson MC, Saczynski JS, Rebok GW, Seeman T, Glass TA, McGill S, Tielsch J, Frick KD, Hill J, Fried LP. Exploring the effects of an "everyday" activity program on executive function and memory in older adults: Experience Corps. Gerontologist. 2008 Dec;48(6):793-801. doi: 10.1093/geront/48.6.793. PMID 19139252
- [Background] Glass TA, Freedman M, Carlson MC, Hill J, Frick KD, Ialongo N, McGill S, Rebok GW, Seeman T, Tielsch JM, Wasik BA, Zeger S, Fried LP. Experience Corps: design of an intergenerational program to boost social capital and promote the health of an aging society. J Urban Health. 2004 Mar;81(1):94-105. doi: 10.1093/jurban/jth096. PMID 15047788
- [Background] Rebok GW, Carlson MC, Glass TA, McGill S, Hill J, Wasik BA, Ialongo N, Frick KD, Fried LP, Rasmussen MD. Short-term impact of Experience Corps participation on children and schools: results from a pilot randomized trial. J Urban Health. 2004 Mar;81(1):79-93. doi: 10.1093/jurban/jth095. PMID 15047787
- [Derived] Varma VR, Tan EJ, Gross AL, Harris G, Romani W, Fried LP, Rebok GW, Carlson MC. Effect of Community Volunteering on Physical Activity: A Randomized Controlled Trial. Am J Prev Med. 2016 Jan;50(1):106-110. doi: 10.1016/j.amepre.2015.06.015. Epub 2015 Sep 2. PMID 26340864